CLINICAL TRIAL: NCT02895061
Title: Effectiveness Between Daily Versus Pulse Oral Alfacalcidol for Secondary Hyperparathyroidism in Chronic Hemodialysis Patients: A Randomized Controlled Trial and Multicenter Study
Brief Title: Effectiveness of Oral Alfacalcidol for Secondary Hyperparathyroidism in Chronic Hemodialysis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PMK-0007
Record Dates: First submitted 2016-09-04; First posted 2016-09-09 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2015-01

CONDITIONS: Alfacalcidol, Secondary Hyperparathyroidism, Hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — alfacalcidol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Daily (Experimental): A: oral daily alfacalcidol treatments total 6 microgram/week
  Interventions: Drug: Alfacalcidol
- B: Pulse (Experimental): B: pulse (trice a week) alfacalcidol treatments total 6 microgram/week
  Interventions: Drug: Alfacalcidol

INTERVENTIONS:
Drug: Alfacalcidol — Alfacalcidol 1 microgram/capsule
  Other Names: oral daily alfacalcidol treatments total 6 microgram/week

SUMMARY:
Primary objective was to evaluate the efficacy between daily and pulse oral alfacalcidol treatment of SHPT in chronic hemodialysis patients, a 12-week treatment. Secondary objective was to observe the adverse effects between these two treatment regimens.

DETAILED DESCRIPTION:
ESRD patients with secondary hyperparathyroidism in 3 hemodialysis centers were enrolled. They were assigned to either oral daily or pulse (trice a week) alfacalcidol treatments using block-of-4 randomization. Alfacalcidol in both groups were equal at the dose of 6 microgram per week. Clinical and laboratory data were obtained at baseline and were monitored every 4 weeks for 12 weeks. Primary outcome was the difference of the mean PTH reduction between two groups at the end of the study by unpaired-T test. All possible adverse events were carefully monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 y ESRD on HD KT/V ≥ 3.6/wk 2˚HPT Stable in P binder for 4 wk

Exclusion Criteria:

* Alfacalcidol allergy Serum Ca ≥ 10.5 mg/dL Serum P ≥ 5.5 mg/dL Pregnancy On phenytoin, phenobarbital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome was the difference of the mean PTH reduction between two groups at the end of the study by unpaired-T test. | 12 week
  mean PTH reduction between two groups at the end of the study by unpaired-T test.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gu Y, Ding F, Chen N, Mei CL, Qian JQ, Wang XY, Shi W, Hou FF, Li XW, Wang M, Chen YP. Comparisons between oral pulse alfacalcidol therapy and daily therapy in maintenance hemodialysis patients with secondary hyperparathyroidism: a randomized, controlled, and multicenter study. Ren Fail. 2005;27(2):205-12. PMID 15807187
- [Result] Tarrass F, Yazidi A, Sif H, Zamd M, Benghanem MG, Ramdani B. A randomized trial of intermittent versus continuous oral alfacalcidol treatment of hyperparathyroidism in end-stage renal disease. Clin Nephrol. 2006 Jun;65(6):415-8. doi: 10.5414/cnp65415. PMID 16792136
- [Result] Llach F, Yudd M. Pathogenic, clinical, and therapeutic aspects of secondary hyperparathyroidism in chronic renal failure. Am J Kidney Dis. 1998 Oct;32(2 Suppl 2):S3-12. doi: 10.1053/ajkd.1998.v32.pm9808139. No abstract available.